CLINICAL TRIAL: NCT07209891
Title: COMPARISON STUY OF KINESIOTAPE AND LOW-LEVEL LASER THERAPY ON HYPERTROPHIC SCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Huda Badr Abd El Hamed, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: National institute of laser
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Hypertrophic Scar; Burn Scar (Post-burn); Burns
Keywords: Hypertrophic Scar; Burn; Kinesio Taping; VAS; Schiotz Tonometer; Photobiomodulation.; Low-Level Laser Therapy
MeSH Terms: conditions — Cicatrix, Hypertrophic; Burns | interventions — Athletic Tape; Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Sixty male and female patients with post-burn hypertrophic scars, aged 10-30years, participated in this randomized controlled trial. Patients were randomly assigned to three equal groups: Group A received kinesio tape and medication, Group B received low level laser therapy and medication, and Group C received kinesio tape and low-level laser therapy
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- kinesio tape (Experimental): Kinesiotape was used to cover the full extent of the scar tissue
  Interventions: Device: Kinesio Tape; Other: Standardized Scar Care (concomitant for all arms)
- low-level laser (Experimental): Giotto MED SPA-Italy-Ga-As low-level laser with the following parameters: wavelength 905 nm, energy density 16.2 J/cm2, pulsed mode with frequency 3000 Hz, and max output power 30 W. The application technique was a circular cluster probe with three output beams that each produced 30 W of power. The length of therapy varies according on the size of the scar.
  Interventions: Device: Low-Level Laser Therapy (LLLT), 905-nm pulsed Ga-As; Other: Standardized Scar Care (concomitant for all arms)
- kinesio tape and lowlevel laser (Experimental): combined treatment of low-level laser and kinesio tape
  Interventions: Device: Kinesio Tape; Device: Low-Level Laser Therapy (LLLT), 905-nm pulsed Ga-As; Other: Standardized Scar Care (concomitant for all arms)

INTERVENTIONS:
Device: Kinesio Tape — Cotton elastic tape applied along the full length/width of the target hypertrophic scar with ~25-50% stretch while the scar is on gentle lengthening. Continuous wear; replaced every 2-3 days.
  Arms: kinesio tape; kinesio tape and lowlevel laser
Device: Low-Level Laser Therapy (LLLT), 905-nm pulsed Ga-As — Fluence 16.2 J/cm² at skin; pulse frequency 3000 Hz; session duration ~15 min at standardized distance (~10 cm) using an orange medical filter; protective eyewear for patient and staff.
  Arms: kinesio tape and lowlevel laser; low-level laser
Other: Standardized Scar Care (concomitant for all arms) — Uniform background care applied across all groups; recorded in CRFs; prohibited co-interventions (e.g., intralesional steroids, microneedling, ablative lasers, new pressure garments during the study).

SUMMARY:
Hypertrophic scars after burn injury often cause pain, stiffness, and cosmetic concerns. Kinesio taping (KT) and low-level laser therapy (LLLT; photobiomodulation) are widely used, yet direct comparisons and combined-therapy data remain limited. This single-center, three-arm, parallel randomized controlled trial will compare KT alone, LLLT alone, and their combination in patients with post-burn hypertrophic scars. Sixty participants will be randomized (1:1:1) to receive KT (reapplied every 2-3 days), LLLT using a 905-nm pulsed device (three sessions per week), or KT+LLLT for 8 weeks; all groups receive standardized scar care. Outcome assessors will be blinded. The primary outcome is change in scar pliability/firmness measured with a modified Schiotz tonometer from baseline to week 8. Secondary outcomes include change in pain intensity on a 10-cm visual analogue scale and treatment-related adverse events; an optional assessment at week 12 will evaluate durability. We hypothesize that KT+LLLT will produce greater improvements in elasticity and pain than either modality alone. The trial will be conducted at the Faculty of Physical Therapy, Cairo University (Giza, Egypt). Sponsor: Cairo University; Collaborators: National Institute of Laser Enhanced Sciences (NILES) and Faculty of Physical Therapy.

DETAILED DESCRIPTION:
Objective: Compare the effects of kinesio taping (KT), low-level laser therapy (LLLT), and their combination on pliability and pain of post-burn hypertrophic scars.

Design: Single-center, three-arm, parallel randomized controlled trial (1:1:1); assessor- and analyst-blinded.

Setting: Outpatient clinic, Faculty of Physical Therapy, Cairo University (Giza, Egypt).

Participants: ~60 patients with clinically diagnosed hypertrophic scars after burns; able to complete 8-week treatment; standard exclusions for open wounds, infection, photosensitivity, etc.

Interventions:

Arm A: KT + standardized scar care (tape reapplied every 2-3 days).

Arm B: LLLT (905-nm pulsed device; ~16.2 J/cm²; 3×/week).

Arm C: KT + LLLT on the same schedule.

Duration: 8-week treatment; optional week-12 follow-up for durability.

Primary Outcome: Change in scar pliability/firmness (modified Schiotz tonometer) from baseline to week 8.

Secondary Outcomes: Change in pain (10-cm VAS); treatment-related adverse events; optional week-12 persistence.

Randomization/Concealment: Computer-generated sequence; SNOSE envelopes.

Analysis: Intention-to-treat; linear mixed-effects models with adjusted pairwise contrasts (Holm/Bonferroni).

Sponsor: Cairo University. Collaborators: National Institute of Laser Enhanced Sciences (NILES) and Faculty of Physical Therapy, Cairo University.

Hypothesis: KT+LLLT will yield greater improvements than either modality alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 10 and 30 years. Presence of clinically diagnosed hypertrophic scars secondary to burn injuries, occurring between two months and four years after complete wound healing No history of other systemic or local pathologies that could affect scar characteristics or response to treatment. Ability and willingness to comply with the treatment protocol and attend all scheduled sessions

Exclusion Criteria:

* Open wounds or ulceration at or near the scarred area. Systemic medical conditions such as uncontrolled diabetes mellitus, cardiovascular disease, or a history of skin malignancy in the treatment region. Diagnosed deep vein thrombosis (DVT).Non-adherence, unwillingness to participate, or inability to follow the protocol. Cognitive impairment, psychiatric illness, or communication barriers affecting informed consent or participation.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Schiotz Tonometer | Baseline (Week 0) ,Week 8.
  The Riester Schiotz tonometer is used as an objective tool to assess hypertrophic scar elasticity The device displayed readings on a scale from 0 to 20. Indentation values were then converted to millimeters of mercury (mmHg) using a standardized conversion chart provided with the device

SECONDARY OUTCOMES:
2. Pain Assessment by Visual Analogue Scale (VAS) | Baseline (Week 0) , Week 8.
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100

CONTACTS AND LOCATIONS:
Locations (1):
- Huda Badr Abd Elhamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR